CLINICAL TRIAL: NCT01192659
Title: Identification of Risk Factors for Low Lymphocyte Count in Patients With Type 2 Diabetes: An Analysis of Data From the SAVOR Study
Brief Title: Risk Factors for Low Lymphocyte Count in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV181-102
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients treated with saxagliptin or placebo: Patients will be treated with saxagliptin or placebo, on top of whatever baseline treatment for diabetes the patient is already receiving.
- Patients currently or previously on treatment: Patients currently or previously on (within 6 months) treatment with DPP4 inhibitors and/or GLP-1 mimetics are excluded.

SUMMARY:
The purpose of this study is to identify risk factors for low lymphocyte count among patients with type 2 diabetes who are treated with oral antidiabetic drugs.

DETAILED DESCRIPTION:
Involving a secondary analysis of data collected prospectively from a defined cohort, for the SAVOR trial.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in SAVOR
* Diagnosed with T2DM
* Baseline HbA1c ≥6.5% (based on the last measured and documented laboratory measurement within 6 months)
* Age 40 or older
* High risk for a cardiovascular event

Exclusion Criteria:

* Not enrolled in SAVOR
* Current or previous treatment with DPP4 inhibitors and/or GLP-1 or incretin mimetics.
* Acute vascular event
* Pregnancy
* HIV/AIDS
* Severe autoimmune disease
* Current chronic steroid use

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the Saxagliptin Assessment of Vascular Outcomes Recorded in Diabetes Mellitus study, which is a randomized, placebo-controlled phase 4 study of cardiovascular outcomes). 12,000 patients with type 2 diabetes and either a history of a cardiovascular event or multiple risk factors for vascular disease. Patients will be distributed as follows: at least 30% in North America, approximately 30% in Europe, and the remainder in South America, Asia, Australia, and South Africa.
Sampling Method: Non-Probability Sample
Enrollment: 16492 (Actual)
Dates: Start 2010-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To identify risk factors for lymphopenia, defined as an absolute lymphocyte count < 500 cells/μl, or investigator reported lymphopenia, in the SAVOR study population. | 60 months

SECONDARY OUTCOMES:
To identify risk factors for absolute lymphocyte count <750 cells/µl or investigator reported lymphopenia. | 60 months
To identify risk factors for decreased lymphocyte count (>=30% decrease from baseline. | 60 months
To evaluate whether risk factors for low lymphocyte counts or decreasing lymphocyte count differ between saxagliptin users and non-users. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4124&filename=CV181-102_Final_Study_Report%20_Redacted.pdf